CLINICAL TRIAL: NCT04161183
Title: Extracoporeal Shock Wave Therapy (ESWT) for the Treatment of Detrusor Underactivity/ Underactive Bladder (DU/UAB) - a Single Center, Randomized, Double-blind, Placebo-controlled, Prospective Study
Brief Title: Extracoporeal Shock Wave Therapy (ESWT) for the Treatment of Detrusor Underactivity/ Underactive Bladder (DU/UAB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201900500A0
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-03

CONDITIONS: Detrusor, Underactive; Detrusor Underactivity
Keywords: shock wave; detrusor underactivity; underactive bladder
MeSH Terms: conditions — Urinary Bladder, Underactive

STUDY DESIGN:
Intervention Model Description: Double blind, placebo control study. Eligible patients will be assigned a randomization number in sequential order and each of the randomization will determine the allocation of one of the two treatment groups (ESWT and Placebo) in 1: 1 ratio as shown below. The ESWT and placebo will be controlled by a research assistance who will not evaluate the therapeutic outcome to ensure the double-blind method.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo treatment (shock wave probe w/o energy)
  Interventions: Device: Placebo
- Extracoporeal shock wave therapy (Experimental): Extracoporeal shock wave therapy (shock wave probe w/ energy)
  Interventions: Device: Extracoporeal shock wave therapy

INTERVENTIONS:
Device: Extracoporeal shock wave therapy — Probe be transcutaneous applied to the region of bladder dome, right upper lateral wall, right lower lateral wall, left upper lateral wall, and left lower lateral wall with 2500 shocks, frequency of 4 pulses per second and maximum total energy flow density 0.25 millijoule/mm2 once a week for 6 weeks
  Arms: Extracoporeal shock wave therapy
Device: Placebo — Probe be transcutaneous applied to the region of bladder dome, right upper lateral wall, right lower lateral wall, left upper lateral wall, and left lower lateral wall with 2500 shocks, frequency of 4 pulses per second but no energy once a week for 6 weeks
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of ESWT for the treatment of patients with DU/UAB

DETAILED DESCRIPTION:
The prevalence of detrusor underactivity/ underactive bladder (DU/UAB) increased with age, which is 9-28% in young men (<50 years), and is up to 48% in the elderly men (>70 years) with non-neurogenic lower urinary tract symptoms. In women aged >70 years, the prevalence of DU ranged from 12% to 45%. Currently, there is a lack of effective pharmacological or surgical treatment of DU/UAB. Previously we demonstrated that extracoporeal shock wave therapy (ESWT) was able to mediate a partial recovery in the contractility of cryoinjury induced DU/UAB model in rats. Wang et al. reported the therapeutic effect of ESWT in the streptozotocin induced diabetic underactive bladder rat model with significantly improved voiding function, enhanced detrusor contractility, increased muscle actin expression and muscle proportion of the bladder wall, and recovery of neuronal integrity and innervations. Taken together, these findings suggest that a potential clinical benefit of ESWT treatment for patients with DU/UAB.

A total of 60 patients with DU/UAB will be enrolled to receive ESWT once a week for 6 weeks or placebo treatment. Patients with DU/UAB symptoms with post void residual (PVR) ≥ 100 mL and proven of DU/UAB without bladder outlet obstruction (BOO) by urodynamic study. Patients should not have uncontrolled acute urinary tract infection, and should not have treated with an investigational device, drug, or procedure for UAB within the last 3 months. Retreatment with ESWT at 3 months if patient reports ineffective will be allowed.

Primary end-point is the change of PVR volume (mL) from baseline to 1 month after treatment. Secondary endpoints include daily frequency, nocturia and FBC as record in 3-day voiding diary, Qmax, Pdet@Qmax, voided volume, PVR and global response assessment (GRA). One visit is required at baseline screening (before first treatment), treatment 1 (V1), treatment 2 (V2), treatment 3 (V3), treatment 4 (V4), treatment 5 (V5), treatment 6 (V6) and 1 month post V6 treatment (V7, primary end-point), and 3 months post V6 treatment (V8). Urine samples will be collected at each time-point for NGF and cytokines tests. Cystoscopy bladder biopsy will be performed at baseline and at 3 months post treatment, optional.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female, at least 20 years of age.
2. History of UAB (defined as bothersome chronic incomplete bladder emptying) for at least 3 months documented in the medical record with recurring UAB symptoms.
3. No UAB symptom relief (unresponsiveness) with previous used medications and/or other treatments.
4. Voiding difficulty (complains of difficulty emptying the bladder).
5. UAB consistent with diabetes, MS, Parkinson's disease, or aging idiopathic.
6. Post void residual ≥ 100 mL.
7. Bladder capacity > 200 mL and < 800 mL.
8. Pressure flow Urodynamic testing demonstrating impaired detrusor contractility or areflexia without evidence of BOO, with maximum detrusor pressure Pdet at Qmax (Pdet@Qmax) of < 20 cmH2O and Maximum flow rate (Qmax) < 15 mL/sec for female, and BCI < 100 and BOOI < 40 for male.
9. Total UAB Questionnaire Score ≥ 3.
10. Females of child-bearing potential agree to use reliable birth control for the entire study duration.
11. Willing and capable of understanding and complying with all requirements of the protocol, including proper completion of the voiding diaries and self-administered questionnaires.
12. Free of active urinary tract infection.
13. Free of bladder outlet obstruction on enrollment.
14. Patient or his/her legally acceptable representative has signed the written informed consent form.
15. Subject on clean intermittent catheterization (CIC) should have been on CIC for at least 1 month and should be able to void spontaneously and not be completely dependent on CIC.

Exclusion Criteria:

1. Female patients who is pregnant, lactating, plans to become pregnant, or with child-bearing potential without contraception.
2. Simultaneously participating in another investigational drug or device study or use of any investigational drug(s) or therapeutic device(s) within 3 months preceding enrollment
3. Has been treated with an investigational device, drug, or procedure for UAB within the last 3 months.
4. History of cancer in pelvic organs, ureters, or kidneys or any cancer that has undergone treatment within the past 12 months.
5. Medical condition or disorder that may limit life expectancy or that may cause protocol deviations (e.g. unable to perform self-evaluations/accurately report medical history, and/or urinary symptoms).
6. History of spinal cord injury affecting urinary function.
7. Patients with uncontrolled acute urinary tract infection. An active urinary tract infection as evidenced by positive urine culture at the time of baseline assessment. If a UTI is confirmed in the baseline sample (e.g., positive urine culture containing > 100,000 cfu/mL in midstream urine), the run-in period should be stopped. After successful treatment of the UTI, the patient can be rescreened and if eligible enroll in the study. If the patient has asymptomatic bacteriuria (i.e., a positive urine culture without clinical signs and symptoms of a UTI), the patient should not be excluded.
8. Currently taking medication(s) that may affect urination, including prescription drugs (i.e. anticholinergics, tricyclic antidepressants, bethanechol), over the counter drugs, dietary and/or herbal supplements, adrenergic antagonists. Alpha adrenergic blockers are allowed to use in a stable condition (longer than 1 month and keeping use during the study period).
9. Pelvic organ prolapses beyond the introitus (e.g., cystocele, rectocele).
10. Prior mesh surgery for stress urinary incontinence or pelvic prolapse.
11. Any other condition which per investigators' judgement, may affect the patient's safety (e.g. significant cardiovascular disease, asthma or other breathing disorders).
12. Patients with bladder outlet obstruction on enrollment.
13. Patients with any contraindication to be urethral catheterization during diagnostic test or treatment or follow-up period.
14. Patients have laboratory abnormalities at screening including:

    ALT > 3 x upper limit of normal range AST > 3 x upper limit of normal range Serum creatinine level > 2 x upper limit of normal range.
15. Patients with any other serious disease considered by the investigator not in the condition to enter the trial.
16. Patients with cortisone treatment 6 week before first LESW therapy.

Other single item of Lab examination also can be retested per Investigator's discretion if abnormality. Patient will be rescreened and randomized into the study once confirmed eligible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Net changes of the mean post void residual (PVR) volume (mL) from baseline to 1 month after the last treatment day | Baseline and 1 month
  Net changes of the PVR from baseline to 1 month after the last treatment day (higher PVR volumes represent a worse outcome)

SECONDARY OUTCOMES:
Net changes of the functional bladder capacity (FBC) as assessed by the maximum urine volume (milliliters) as recorded in 3-day voiding diary | Baseline and 1 month
  Net changes of the functional bladder capacity (FBC) from baseline to 1 month after the last treatment day (higher FBC volumes represent a better outcome)
Net changes of the Global response assessment (GRA) | Baseline and 1 month
  Global response assessment (GRA) of therapeutic result by the patient (categorized from -3 to +3, indicating markedly worse to markedly improved) at 1 month after the last treatment day
Net changes of the maximum flow rate | Baseline and 1 month
  Net changes of the maximum flow rate from baseline to 1 month after the last treatment day (higher maximum flow rate represent a better outcome)
Net changes of the voided volume | Baseline and 1 month
  Net changes of the voided volume from baseline to 1 month after the last treatment day (higher voided volumes represent a better outcome)
Net changes of the Pdet@Qmax | Baseline and 1 month
  Net changes of the Pdet@Qmax from baseline to 1 month after the last treatment day
Net changes of the postvoid residual volume | Baseline and 1 month
  Net changes of the postvoid residual volume from baseline to 1 month after the last treatment day (lower postvoid residual volume represent a better outcome)
Changes of the Underactive Bladder Questionnaire (UAB-Q) score | Baseline and 1 month
  Changes of the UAB-Q score from baseline to 1 month after the last treatment day (lower UAB-Q score represent a better outcome)
Changes of urinary nerve growth factor and cytokines level | Baseline and 1 month
  Changes of the urinary nerve growth factor and cytokines level from baseline to 1 month after the last treatment day

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Tang Hsieh, MD, Study Chair — Institutional Review Board Chang Gung Medical Foundation
Locations (1):
- Chang Gung Memorial Hospital, Chang Gung University College of Medicine, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Miyazato M, Yoshimura N, Chancellor MB. The other bladder syndrome: underactive bladder. Rev Urol. 2013;15(1):11-22. PMID 23671401
- [Background] Chuang YC, Plata M, Lamb LE, Chancellor MB. Underactive Bladder in Older Adults. Clin Geriatr Med. 2015 Nov;31(4):523-33. doi: 10.1016/j.cger.2015.06.002. Epub 2015 Jul 26. PMID 26476113
- [Background] Osman NI, Chapple CR, Abrams P, Dmochowski R, Haab F, Nitti V, Koelbl H, van Kerrebroeck P, Wein AJ. Detrusor underactivity and the underactive bladder: a new clinical entity? A review of current terminology, definitions, epidemiology, aetiology, and diagnosis. Eur Urol. 2014 Feb;65(2):389-98. doi: 10.1016/j.eururo.2013.10.015. Epub 2013 Oct 26. PMID 24184024
- [Background] Brierly RD, Hindley RG, McLarty E, Harding DM, Thomas PJ. A prospective controlled quantitative study of ultrastructural changes in the underactive detrusor. J Urol. 2003 Apr;169(4):1374-8. doi: 10.1097/01.ju.0000055781.07630.aa. PMID 12629365
- [Background] Elbadawi A, Yalla SV, Resnick NM. Structural basis of geriatric voiding dysfunction. II. Aging detrusor: normal versus impaired contractility. J Urol. 1993 Nov;150(5 Pt 2):1657-67. doi: 10.1016/s0022-5347(17)35867-6. PMID 8411454
- [Background] Jiang YH, Kuo HC. Urothelial Barrier Deficits, Suburothelial Inflammation and Altered Sensory Protein Expression in Detrusor Underactivity. J Urol. 2017 Jan;197(1):197-203. doi: 10.1016/j.juro.2016.07.071. Epub 2016 Jul 17. PMID 27436428
- [Background] Cho KJ, Koh JS, Choi J, Kim JC. Changes in Adenosine Triphosphate and Nitric Oxide in the Urothelium of Patients with Benign Prostatic Hyperplasia and Detrusor Underactivity. J Urol. 2017 Dec;198(6):1392-1396. doi: 10.1016/j.juro.2017.06.080. Epub 2017 Jun 24. PMID 28655527
- [Background] Andersson KE. Detrusor underactivity/underactive bladder: new research initiatives needed. J Urol. 2010 Nov;184(5):1829-30. doi: 10.1016/j.juro.2010.08.048. Epub 2010 Sep 17. No abstract available. PMID 20846686
- [Background] Osman NI, Esperto F, Chapple CR. Detrusor Underactivity and the Underactive Bladder: A Systematic Review of Preclinical and Clinical Studies. Eur Urol. 2018 Nov;74(5):633-643. doi: 10.1016/j.eururo.2018.07.037. Epub 2018 Aug 20. PMID 30139634
- [Background] Wang HJ, Cheng JH, Chuang YC. Potential applications of low-energy shock waves in functional urology. Int J Urol. 2017 Aug;24(8):573-581. doi: 10.1111/iju.13403. Epub 2017 Jul 11. PMID 28697536
- [Background] Chuang YC, Tyagi P, Wang HJ, Huang CC, Lin CC, Chancellor MB. Urodynamic and molecular characteristics of detrusor underactivity in a rat cryoinjury model and effects of low energy shock wave therapy. Neurourol Urodyn. 2018 Feb;37(2):708-715. doi: 10.1002/nau.23381. Epub 2017 Aug 2. PMID 28767169
- [Background] Chuang YC, Tyagi P, Luo HL, Lee WC, Wang HJ, Huang CC, Chancellor MB. Long-term functional change of cryoinjury-induced detrusor underactivity and effects of extracorporeal shock wave therapy in a rat model. Int Urol Nephrol. 2019 Apr;51(4):617-626. doi: 10.1007/s11255-019-02095-4. Epub 2019 Feb 22. PMID 30796726
- [Background] Wang HS, Oh BS, Wang B, Ruan Y, Zhou J, Banie L, Lee YC, Tamaddon A, Zhou T, Wang G, Lin G, Lue TF. Low-intensity extracorporeal shockwave therapy ameliorates diabetic underactive bladder in streptozotocin-induced diabetic rats. BJU Int. 2018 Sep;122(3):490-500. doi: 10.1111/bju.14216. Epub 2018 Apr 20. PMID 29603534
- [Background] Zissler A, Steinbacher P, Zimmermann R, Pittner S, Stoiber W, Bathke AC, Sanger AM. Extracorporeal Shock Wave Therapy Accelerates Regeneration After Acute Skeletal Muscle Injury. Am J Sports Med. 2017 Mar;45(3):676-684. doi: 10.1177/0363546516668622. Epub 2016 Oct 13. PMID 27729321
- [Background] Wang B, Zhou J, Banie L, Reed-Maldonado AB, Ning H, Lu Z, Ruan Y, Zhou T, Wang HS, Oh BS, Wang G, Qi SL, Lin G, Lue TF. Low-intensity extracorporeal shock wave therapy promotes myogenesis through PERK/ATF4 pathway. Neurourol Urodyn. 2018 Feb;37(2):699-707. doi: 10.1002/nau.23380. Epub 2017 Aug 1. PMID 28763567
- [Background] Uren AD, Cotterill N, Harding C, Hillary C, Chapple C, Klaver M, Bongaerts D, Hakimi Z, Abrams P. Qualitative Exploration of the Patient Experience of Underactive Bladder. Eur Urol. 2017 Sep;72(3):402-407. doi: 10.1016/j.eururo.2017.03.045. Epub 2017 Apr 8. PMID 28400168
- [Background] Zimmermann R, Cumpanas A, Miclea F, Janetschek G. Extracorporeal shock wave therapy for the treatment of chronic pelvic pain syndrome in males: a randomised, double-blind, placebo-controlled study. Eur Urol. 2009 Sep;56(3):418-24. doi: 10.1016/j.eururo.2009.03.043. Epub 2009 Mar 25. PMID 19372000
- See also: Astellas Pharma Inc (Astellas Pharma Europe B.V.). A Study of ASP8302 in Participants With Underactive Bladder. ClinicalTrials.gov Identifier: NCT03702777 — https://clinicaltrials.gov/ct2/show/NCT03702777?term=NCT03702777&draw=2&rank=1

DOCUMENTS (2):
  • Study Protocol (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT04161183/Prot_002.pdf
  • Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT04161183/SAP_003.pdf